CLINICAL TRIAL: NCT03807271
Title: Computer-assisted Anaesthesia Using Pharmacokinetic/Pharmacodynamic Model
Brief Title: Calculated and Graphically Produced Depth of Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018/2176
Record Dates: First submitted 2019-01-09; First posted 2019-01-16 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Anesthesia, General
Keywords: Anesthesia, Methods; Anesthesia, Analysis; Patient Safety; Anesthetics/administration and dosage

STUDY DESIGN:
Who Masked: Participant
Masking Description: The anesthesia team must know if the anesthesia will be given by standard procedure or guided by the calculating device in addition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart Pilot(R) View (Experimental): Anesthesia provided by standard procedure, additionally guided by Smart Pilot(R) View, a device with calculated and graphically produced depth of anesthesia.
  Interventions: Device: Calculated and graphically produced depth of anesthesia (Smart Pilot® View)
- Standard (No Intervention): Anesthesia provided by standard procedure.

INTERVENTIONS:
Device: Calculated and graphically produced depth of anesthesia (Smart Pilot® View) — Smart Pilot® View is a device integrated in the ventilator used under general anesthesia. The depth of anesthesia is calculated based on age, weight, height and the medication given - both volatiles and intravenous. The device does not control the supply of medication directly, but provides an estimate of anesthesia depth that can help the anesthesia team to control the supply of anesthetic agents under general anesthesia, ie indirectly.
  Arms: Smart Pilot(R) View

SUMMARY:
There are studies that suggest that unsatisfying levels of anesthesia can cause peri- and postoperative complications in the patient undergoing surgery. Having a unnecessary "deep" anesthesia level can be harmful, causing acute renal failure, injure to myocard, cause delirium and increase the mortality rate. Being too "light", on the other hand, can make the patient experience awareness when muscle relaxant is used. This can lead to serious psychological struggles.

Evaluating the depth of anesthesia is the most important task of the anesthesia team, but can be difficult because clinical signs depend on many factors. In addition to clinical evaluation, EEG is commonly used for interpreting the level of anesthesia in todays practice. Unfortunately, this method is not always accurate and has a delay.

New devices are now developed to calculate the anesthesia level based on the drugs given. The level is simultaneously presented graphically on screen. The purpose of this study is to investigate and compare clinical parameters within patients undergoing general anesthesia, with and without the use of such devices. Hemodynamic stability, less use of adrenergics, higher EEG-levels, a more rapid wake-up and shorter time in post operative care can indicate a more precise level of anesthesia, hence, promote patient safety.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* Standard premedication
* General anesthesia, total intravenous anesthesia

Exclusion Criteria:

* Alcoholics
* BMI 35 or higher
* Unable to give consent

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Mean Arterial Pressure (MAP) | Maximum 5 hours

SECONDARY OUTCOMES:
Heart Rate (HR) | Maximum 5 hours
Bispectral Index (BIS) | Maximum 5 hours
Total dosis of Propofol in milligrams | Maximum 5 hours
Total dosis of Remifentanil in micrograms | Maximum 5 hours
Total dosis of Ephedrine in milligrams | Maximum 5 hours
Total dosis of Phenylephrine in micrograms | Maximum 5 hours
Total dosis of Atropine in micrograms | Maximum 5 hours
Total dosis of Norepinephrine in micrograms | Maximum 5 hours
Duration of surgery in minutes | Maximum 5 hours
Duration of anesthesia in minutes | Maximum 5 hours
Time until extubation in minutes | Maximum 5 hours
Duration of stay in postoperative ward in minutes | Maximum 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Vifladt, MD, Study Director — Norwegian University of Science and Technology
Locations (1):
- Anestesiavdeling Lillehammer Sykehus, Lillehammer, Oppland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strand H, Elshaug AC, Bernersen O, Ballangrud R. Effectiveness of the advisory display SmartPilot(R) view in the assessment of anesthetic depth in low risk gynecological surgery patients: a randomized controlled trial. BMC Anesthesiol. 2022 Feb 28;22(1):57. doi: 10.1186/s12871-022-01593-w. PMID 35227197